CLINICAL TRIAL: NCT02792829
Title: A Randomized Three-Arm, Single-dose, Two-period Crossover Study to Evaluate the Relative Bioavailability and Palatability of a Lenvatinib Suspension Compared to the Capsule Formulation in Adult Healthy Volunteers
Brief Title: Crossover Study to Evaluate the Relative Bioavailability and Palatability of a Lenvatinib Suspension Compared to the Capsule Formulation in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-009
Record Dates: First submitted 2015-10-15; First posted 2016-06-08 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability of Lenvatinib suspension; Palatability of Lenvatinib suspension; Lenvatinib; Lenvima; E7080; Capsule formulation; Healthy volunteers
MeSH Terms: interventions — lenvatinib

ARMS (3):
- Lenvatinib 11 mg (suspension formulation) (Experimental): Arm 1 will have 2 sequences:
  1. Sequence 1 - Treatment Period 1: 11 mg suspension (2 capsules, 1 x 10 mg and 1 x 1 mg); Treatment Period 2: 11 mg capsules (2 capsules, 1 x 10 mg and 1 x 1 mg)
  2. Sequence 2 - Treatment Period 1: 11 mg capsules (2 capsules, 1 x 10 mg and 1 x 1 mg); Treatment Period 2: 11 mg suspension (2 capsules, 1 x 10 mg and 1 x 1 mg)
  Interventions: Drug: Lenvatinib
- Lenvatinib 11 mg (2 vs 5 capsules) (Experimental): Arm 2 will have 4 sequences:
  1. Sequence 3 - Treatment Period 1: 11 mg suspension (5 capsules, 2 x 4 mg and 3 x 1 mg) WATER; Treatment Period 2: 11 mg suspension (2 capsules, 1 x 10 mg and 1 x 1 mg) APPLE JUICE
  2. Sequence 4 - Treatment Period 1: 11 mg suspension (5 capsules, 2 x 4 mg and 3 x 1 mg capsules) APPLE JUICE; Treatment Period 2: 11 mg suspension (2 capsules, 1 x 10 mg and 1 x 1 mg capsules) WATER
  3. Sequence 5 - Treatment Period 1: 11 mg suspension (2 capsules, 1 x 10 mg and 1 x 1 mg capsules) WATER; Treatment Period 2: 11 mg suspension (5 capsules, 2 x 4 mg and 3 x 1 mg capsules) APPLE JUICE
  4. Sequence 6 - Treatment Period 1: 11 mg suspension (2 capsules, 1 x 10 mg and 1 x 1 mg capsules) APPLE JUICE; Treatment Period 2: 11 mg suspension (5 capsules, 2 x 4 mg and 3 x 1 mg capsules) WATER
  Interventions: Drug: Lenvatinib
- Lenvatinib 23 mg (Experimental): Arm 3 will have 2 sequences:
  1. Sequence 7 - Treatment Period 1: 23 mg suspension (5 capsules, 2 x 10 mg and 3 x 1 mg capsules) taken 23 hours after preparation; Treatment Period 2: 23 mg suspension (5 capsules, 2 x 10 mg and 3 x 1 mg capsules) taken 2 hours after preparation
  2. Sequence 8 - Treatment Period 1: 23 mg suspension (5 capsules, 2 x 10 mg and 3 x 1 mg capsules) taken 2 hours after preparation; Treatment Period 2: 23 mg suspension (5 capsules, 2 x 10 mg and 3 x 1 mg capsules) taken 23 hours after preparation
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — All participants will receive one single dose in each of the 2 treatment periods (total of 2 doses). The total duration of the treatment periods is 12 days (6 days per period) in healthy adult volunteers.
  Other Names: Lenvima; E7080

SUMMARY:
The study will be conducted in adult healthy participants and will consist of two phases: Prerandomization and Randomization. The Prerandomization Phase will consist of 2 periods: a Screening Period and a Baseline Period. The Randomization Phase will consist of 2 Periods (each 6 days long) separated by a 1-day long Baseline Period and End of Treatment (EOT) Period. A total of 60 participants will be enrolled into one of three arms. Arms 1 and 3 consist of 2 sequences, and Arm 2 consists of 4 sequences (as this is an incomplete block design with 2 factors [number of capsules and whether water or apple juice is used as vehicle]). Each participant will be randomized into one of 8 sequences.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants age greater than or equal to 18 years and less than or equal to 55 years old at time of informed consent
2. Nonsmokers or smokers who smoke no more than 10 cigarettes per day
3. BMI greater than or equal to 18 and less than or equal to 32 kg/m2 at screening
4. Adequate liver function, defined as: bilirubin less than or equal to 1.5 X the upper limit of normal (ULN), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and alanine aminotransferase (ALT) less than or equal to 1.5 X ULN
5. Adequate renal function defined as creatinine clearance greater than 70 mL/min calculated using the Cockcroft and Gault formula
6. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L, or equivalent units of B-hCG. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
7. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
8. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the participant must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
9. Male participants must have had a successful vasectomy (confirmed azoospermia), or they and their female partners must meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.
10. Provide written informed consent
11. Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Clinically significant illness that requires medical treatment within 8 weeks prior, or a clinically significant infection that requires medical treatment within 4 weeks prior to dosing
2. Evidence of disease that may influence the outcome of the study, within 4 weeks prior to dosing; eg, psychiatric disorders and disorders of the gastrointestinal (GI) tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
3. Any history of surgery that may affect PK profiles of lenvatinib eg, hepatectomy, nephrotomy, digestive organ resection, at screening or baseline
4. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that requires medical treatment at screening or baseline
5. Prolonged QTcF interval (QTcF greater than 450 ms) demonstrated on ECG at screening or baseline
6. Known history of clinically significant drug allergy at Screening or Baseline
7. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
8. Known history of sensitivity to any of the components of the test products
9. Known to be human immunodeficiency virus (HIV) positive at screening
10. Active viral hepatitis (A, B, or C) as demonstrated by positive serology at screening
11. History of drug or alcohol dependency or abuse within the 2 years prior to screening, or those who have a positive urine drug test or breath alcohol test at Screening or Baseline
12. Engagement in strenuous exercise within 2 weeks prior to check-in (eg, marathon runners, weight lifters)
13. Any medical or other condition that would make the participant in the opinion of the investigator or sponsor, unsuitable for the study or who, in the opinion of the investigator, are not likely to complete the study for any reason
14. Intake of herbal preparations containing St. John's Wort within 4 weeks prior to dosing
15. Use of prescription drugs within 4 weeks prior to dosing
16. Intake of over-the-counter (OTC) medications within 2 weeks prior to dosing
17. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week prior to dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Lenvatinib 11 mg: Suspension+ Capsules (CAP): Participants received lenvatinib 11 mg (milligram), suspension in water (prepared using 1 capsule of 10 mg and 1 capsule of 1 mg) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 11 mg, capsules (1 capsules of 10mg and 1 capsules of 1 mg) on Day 8 of Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 1: Lenvatinib 11 mg: CAP+ Suspension: Participants received lenvatinib 11 mg, capsules (1 capsules of 10mg and 1 capsules of 1 mg) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 11 mg, suspension in water (prepared using 1 capsule of 10 mg and 1 capsule of 1 mg) on Day 8 of Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2:Lenvatinib 11mg Suspension:5 CAP-Water+2 Cap-Apple Juice: Participants received lenvatinib 11mg, suspension in water (prepared using 2 capsule of 4 mg each and 3 capsule of 1 mg each) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 11mg, suspension in apple juice (prepared using 1 capsules of 10mg and 1 capsules of 1 mg) on Day 8 of Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2:Lenvatinib 11mg Suspension:5 CAP-Apple Juice+2 CAP-Water: Participants received lenvatinib 11mg, suspension in apple juice (prepared using 2 capsule of 4 mg each and 3 capsule of 1 mg each) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 11mg, suspension in water (prepared using 1 capsule of 10 mg and 1 capsule of 1 mg) on Day 8 of Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2:Lenvatinib 11mg Suspension:2 CAP-Water+5 CAP-Apple Juice: Participants received lenvatinib 11mg, suspension in water (prepared using 1 capsule of 10 mg and 1 capsule of 1 mg) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 11mg, suspension in apple juice (prepared using 2 capsules of 4 mg each and 3 capsules of 1 mg each) on Day 8 of Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2:Lenvatinib 11mg Suspension:2 CAP-Apple Juice+5 CAP-Water: Participants received lenvatinib 11mg, suspension in apple juice (prepared using 1 capsule of 10 mg and 1 capsule of 1 mg) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 11mg, suspension in water (prepared using 2 capsules of 4 mg each and 3 capsules of 1 mg) on Day 8 on Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 3:Lenvatinib 23mg Suspension Taken at:23 Hours+2 Hours: Participants received lenvatinib 11mg, suspension in water taken 23 hours after preparation (prepared using 2 capsules of 10 mg each and 3 capsules of 1 mg of each) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 23mg, suspension in water taken 2 hours after preparation (prepared using 2 capsules of 10 mg each and 3 capsules of 1 mg) on Day 8 of Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 3:Lenvatinib 23mg Suspension Taken at:2 Hours+23 Hours: Participants received lenvatinib 23mg, suspension in water taken 2 hours after preparation (prepared using 2 capsules of 10 mg each and 3 capsules of 1 mg of each) on Day 1 of Treatment Period 1 followed by a 6-days wash-out period, further followed by lenvatinib 23mg, suspension in water taken 23 hours after preparation (prepared using 2 capsules of 10 mg each and 3 capsules of 1 mg) on Day 8 of Treatment Period 2. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
Period: Treatment Period 1
Arm/Group | Arm 1: Lenvatinib 11 mg: Suspension+ Capsules (CAP) | Arm 1: Lenvatinib 11 mg: CAP+ Suspension | Arm 2:Lenvatinib 11mg Suspension:5 CAP-Water+2 Cap-Apple Juice | Arm 2:Lenvatinib 11mg Suspension:5 CAP-Apple Juice+2 CAP-Water | Arm 2:Lenvatinib 11mg Suspension:2 CAP-Water+5 CAP-Apple Juice | Arm 2:Lenvatinib 11mg Suspension:2 CAP-Apple Juice+5 CAP-Water | Arm 3:Lenvatinib 23mg Suspension Taken at:23 Hours+2 Hours | Arm 3:Lenvatinib 23mg Suspension Taken at:2 Hours+23 Hours
Started | 10 | 10 | 5 | 5 | 5 | 5 | 10 | 10
Completed | 10 | 10 | 5 | 5 | 5 | 5 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash Out Period
Arm/Group | Arm 1: Lenvatinib 11 mg: Suspension+ Capsules (CAP) | Arm 1: Lenvatinib 11 mg: CAP+ Suspension | Arm 2:Lenvatinib 11mg Suspension:5 CAP-Water+2 Cap-Apple Juice | Arm 2:Lenvatinib 11mg Suspension:5 CAP-Apple Juice+2 CAP-Water | Arm 2:Lenvatinib 11mg Suspension:2 CAP-Water+5 CAP-Apple Juice | Arm 2:Lenvatinib 11mg Suspension:2 CAP-Apple Juice+5 CAP-Water | Arm 3:Lenvatinib 23mg Suspension Taken at:23 Hours+2 Hours | Arm 3:Lenvatinib 23mg Suspension Taken at:2 Hours+23 Hours
Started | 10 | 10 | 5 | 5 | 5 | 5 | 10 | 10
Completed | 10 | 10 | 5 | 5 | 5 | 5 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Arm 1: Lenvatinib 11 mg: Suspension+ Capsules (CAP) | Arm 1: Lenvatinib 11 mg: CAP+ Suspension | Arm 2:Lenvatinib 11mg Suspension:5 CAP-Water+2 Cap-Apple Juice | Arm 2:Lenvatinib 11mg Suspension:5 CAP-Apple Juice+2 CAP-Water | Arm 2:Lenvatinib 11mg Suspension:2 CAP-Water+5 CAP-Apple Juice | Arm 2:Lenvatinib 11mg Suspension:2 CAP-Apple Juice+5 CAP-Water | Arm 3:Lenvatinib 23mg Suspension Taken at:23 Hours+2 Hours | Arm 3:Lenvatinib 23mg Suspension Taken at:2 Hours+23 Hours
Started | 10 | 10 | 5 | 5 | 5 | 5 | 10 | 10
Completed | 10 | 9 | 5 | 5 | 4 | 5 | 9 | 8
Not Completed | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Not completed — Non compliance with alcohol prohibition | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Use of proscribed medications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Groups:
- Arm 1: 11 mg Lenvatinib Suspension in Water: On the mornings of Days 1 and 8, following an overnight fast of at least 10 hours, participants were administered lenvatinib (11 mg) suspension in water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 1: 11 mg Lenvatinib Capsule With Water: On the administered lenvatinib (11 mg) capsules with 240 mL (8 fluid ounces) of water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Water): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 5 capsules of lenvatinib (11 mg total) in water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Juice): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 5 capsules of lenvatinib (11 mg total) in apple juice. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Water): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 2 capsules of lenvatinib (11 mg total) in water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Juice): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 2 capsules of lenvatinib (11 mg total) in apple juice. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours): On the mornings of Days 1 and 8, following an overnight fast of at least 10 hours, participants were administered lenvatinib (23 mg) suspension in water, which had been prepared 23 hours prior to administration. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours): On the mornings of Days 1 and 8, following an overnight fast of at least 10 hours, participants were administered lenvatinib (23 mg) suspension in water, which had been prepared 2 hours prior to administration. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Total: Total of all reporting groups
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Juice) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours) | Total
Number analyzed (Participants) | 10 | 10 | 5 | 5 | 5 | 5 | 10 | 10 | 60
Age, Customized [Count of Participants; unit: Participants]
  18 to 65 years | 10 | 10 | 5 | 5 | 5 | 5 | 10 | 10 | 60
Sex/Gender, Customized [Number; unit: Participants]
  Male | 9 | 7 | 5 | 3 | 3 | 3 | 5 | 7 | 42
  Female | 1 | 3 | 0 | 2 | 2 | 2 | 5 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC(0-t))
Description: Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance liquid chromatography/tandem mass spectrometry (LC-MS/MS) method using a previously validated assay. The lower limit of quantitation (LLOQ) was 0.25 ng/mL. Plasma pharmacokinetics (PK) data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of AUC(0-t), which were then summarized as the mean and standard deviation for all participants and expressed as hours·nanogram/milliliter (hr·ng/mL).
Time Frame: Treatment Period 1: Day 1 (Visit 2), Day 2 (Visit 3), Days 3 to 6 (Visits 4 to 7); Treatment Period 2: Day 8 (Visit 8), Day 9 (Visit 9), Days 10 to 13 (Visits 10 to 13)
Population: The PK Analysis Set was the group of subjects who had sufficient PK data for at least 1 PK parameter to be derived. Subjects with predose lenvatinib concentration >5% of their own Cmax, and subjects who experienced emesis at or before 2x median tmax were excluded from data analysis for bioavailability.
Measure: Mean (Standard Deviation); unit: hr·ng/mL
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Juice) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
hr·ng/mL | 1330 (452) | 1340 (482) | 1020 (172) | 1500 (706) | 1340 (519) | 1010 (160) | 3010 (919) | 3210 (1040)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Zero to Infinity (AUC(0-inf))
Description: Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates for the AUC(0-inf), which were then summarized as the mean and standard deviation for all participants and expressed as hr·ng/mL.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: hr·ng/mL
Groups:
- Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 5 capsules of lenvatinib (11 mg total) in water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 5 capsules of lenvatinib (11 mg total) in apple juice. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 2 capsules of lenvatinib (11 mg total) in water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 2 capsules of lenvatinib (11 mg total) in apple juice. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours): On the mornings of Days 1 and 8, following an overnight fast of at least 10 hours, participants were administered lenvatinib (23 mg) suspension in water, which had been prepared 23 hours prior to administration. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 17 | 19
hr·ng/mL | 1360 (456) | 1360 (490) | 1040 (177) | 1530 (720) | 1370 (532) | 1030 (161) | 2970 (910) | 3240 (1050)

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC(0-24))
Description: Blood samples were collected during each Treatment Period at predose up to 24 hours post dose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates for the AUC(0-24), which were then summarized as the mean and standard deviation for all participants and expressed as hr·ng/mL.
Time Frame: Treatment Period 1: Predose up to 24 hours post dose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: h·ng/mL
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 8 | 10 | 10 | 18 | 19
h·ng/mL | 1060 (377) | 1050 (383) | 815 (136) | 1150 (564) | 1070 (415) | 804 (136) | 2540 (785) | 2720 (858)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Zero to 72 Hours (AUC(0-72))
Description: Blood samples were collected during each Treatment Period at predose up to 72 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates for the AUC(0-72), which were then summarized as the mean and standard deviation for all participants and expressed as hr·ng/mL.
Time Frame: Treatment Period 1: Predose up to 72 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: hr·ng/mL
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
hr·ng/mL | 1280 (437) | 1290 (466) | 987 (164) | 1430 (668) | 1290 (500) | 971 (152) | 2930 (887) | 3130 (1010)

5. Primary Outcome: Apparent Clearance (CL/F)
Description: Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates for the CL/F, which were then summarized as the mean and standard deviation for all participants and expressed as liters/hour.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 8 | 10 | 10 | 17 | 19
L/hour | 9.34 (4.36) | 9.47 (4.45) | 10.8 (1.73) | 8.70 (3.44) | 9.10 (3.07) | 10.9 (1.61) | 8.46 (2.65) | 7.73 (2.19)

6. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates for the Vz/F, which were then summarized as the mean and standard deviation for all participants and expressed in liters (L).
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 8 | 10 | 10 | 17 | 19
Liters | 301 (159) | 296 (123) | 356 (74.0) | 317 (131) | 312 (122) | 360 (103) | 247 (95.7) | 238 (122)

7. Primary Outcome: Maximum Concentration (Cmax) of Lenvatinib in Plasma
Description: Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of Cmax, which were then summarized as the mean and standard deviation for all participants and expressed as nanograms/milliliter (ng/mL).
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water): Arm 2 group description: On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 2 capsules of lenvatinib (11 mg total) in water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Arm 3: 11 mg Lenvatinib Suspension in Water (2 Hours): On the mornings of Days 1 and 8, following an overnight fast of at least 10 hours, participants were administered lenvatinib (11 mg) suspension in water, which had been prepared 23 hours prior to administration. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 11 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
ng/mL | 133 (52.5) | 126 (44.9) | 115 (22.9) | 150 (65.2) | 138 (61.3) | 105 (21.2) | 358 (128) | 375 (134)

8. Primary Outcome: Time Prior to the First Measureable Concentration of Lenvatinib (Tlag)
Description: Tlag was defined as the time delay between drug administration and the onset of drug absorption. Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of tlag, which were then summarized as the median and full range for all participants and expressed in hours.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
Hours | 0.00 [0.00 to 0.53] | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

9. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of tmax, which were then summarized as the median and full range for all participants and expressed in hours.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
Hours | 3.00 [1.00 to 4.00] | 3.00 [2.00 to 4.00] | 2.52 [2.00 to 3.00] | 3.00 [2.00 to 3.00] | 2.50 [2.00 to 4.00] | 2.00 [2.00 to 3.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 3.00]

10. Primary Outcome: Terminal Elimination Phase Half-life (t1/2)
Description: Blood samples were collected during each Treatment Period at predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose. Plasma concentrations of lenvatinib were quantified by a high-performance LC-MS/MS method using a previously validated assay. The LLOQ was 0.25 ng/mL. Plasma PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of t1/2, which were then summarized as the median and full range for all participants and expressed in hours.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Juice) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
Hours | 22.7 (6.09) | 22.4 (4.67) | 23.2 (5.67) | 25.5 (4.27) | 24.1 (5.05) | 23.1 (6.15) | 20.4 (4.51) | 21.5 (7.35)

11. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Lenvatinib
Description: Safety assessment consisted on monitoring and recording all treatment-emergent adverse events (TEAEs) and SAEs; as well as laboratory evaluations for hematology, blood chemistry, and urine values; periodic measurement of vital signs, electrocardiograms (ECGs); and physical examinations. A TEAE was defined as an adverse events that: 1) emerged during treatment and up to 7 days from the last treatment, having been absent before treatment or at baseline, 2) reemerged during treatment, having been present at Baseline but stopped before treatment, or 3) worsened in severity during treatment relative to the state before treatment, when continuous.
Time Frame: From date of first dose of study treatment to date of last dose of study treatment, up to approximately 2 months 10 days
Population: Safety Analysis Set was the group of subjects who received at least 1 dose of study drug and had at least 1 postdose safety assessment
Measure: Number; unit: Participants
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Juice) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
Participants
  TEAEs | 4 | 6 | 1 | 2 | 4 | 4 | 3 | 4
  Treatment-related TEAEs | 4 | 6 | 0 | 1 | 2 | 1 | 3 | 2
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Summary Scores for Palatability of Lenvatinib
Description: A hedonic Visual Analog Scale (VAS) was used to assess taste likability or "palatability" between a) lenvatinib suspension formulated with water versus the capsule formulation, b) a lenvatinib suspension formulated with with apple juice versus one formulated with water, and c) a lenvatinib suspension formulated with water administered 23 hours versus 2 hours after preparation. All participants selected one face based on flavor, smell, sweetness, acidity, saltiness, bitterness, and texture or mouth feel for each formulation they consumed. Each face had an associated score (1: Very Bad (angry face), 2: Bad (sad face), 3: Maybe Good or Maybe Bad (neutral face), 4: Good (smiling face), 5: Very Good (laughing face)). The VAS hedonic scale scores were summarized using descriptive statistics separately for each arm by formulation (Arm 1), number of capsules (2 vs 5 capsules) and preparation type (water vs apple juice) (Arm 2), and time of administration relative to preparation (Arm 3).
Time Frame: Treatment Period 1, Day 1 (Visit 2); Treatment Period 2, Day 8 (Visit 8)
Population: The Palatability Analysis Set was the group of subjects who received at least 1 dose of study drug and completed the visual analog scale (VAS) in at least one treatment period.
Measure: Median (Full Range); unit: Score on a scale
Groups:
- Lenvatinib 11 mg (Suspension of 5 Capsules in Water): On the mornings of Days 1 and 8 following an overnight fast of at least 10 hours, participants were administered a suspension of 5 capsules of lenvatinib (11 mg total) in water. No food was allowed for at least 4 hours post dose. Water was allowed ad libitum except for the period beginning 1 hour before and until 1 hour after lenvatinib administration. Treatments were administered at the same time on the 2 dosing days. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Lenvatinib 11 mg (Suspension of 5 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 5 Capsules in Juice) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Water) | Arm 2: Lenvatinib 11 mg (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
Number analyzed (Participants) | 19 | 20 | 10 | 9 | 10 | 10 | 18 | 19
Score on a scale
  Flavor Score | 3.0 [1 to 5] | 4.0 [2 to 5] | 3.0 [1 to 5] | 4.0 [2 to 5] | 2.5 [1 to 4] | 4.0 [1 to 5] | 2.0 [1 to 5] | 2.0 [1 to 4]
  Smell Score | 4.0 [3 to 5] | 4.0 [2 to 5] | 3.5 [2 to 5] | 4.0 [3 to 4] | 4.0 [3 to 5] | 4.0 [3 to 5] | 3.0 [1 to 5] | 3.0 [2 to 5]
  Sweetness Score | 3.0 [1 to 5] | 3.0 [1 to 5] | 3.0 [1 to 4] | 4.0 [2 to 5] | 2.0 [1 to 4] | 4.0 [2 to 5] | 2.0 [1 to 4] | 2.0 [1 to 4]
  Acidity Score | 3.0 [1 to 5] | 4.0 [2 to 5] | 3.0 [1 to 5] | 3.0 [2 to 4] | 2.5 [1 to 4] | 4.0 [2 to 5] | 3.0 [1 to 5] | 3.0 [1 to 4]
  Saltiness Score | 3.0 [2 to 5] | 4.0 [1 to 5] | 3.0 [1 to 4] | 4.0 [1 to 5] | 3.0 [2 to 5] | 4.0 [2 to 5] | 3.0 [2 to 5] | 4.0 [1 to 5]
  Bitterness Score | 3.0 [1 to 5] | 3.5 [1 to 5] | 3.0 [1 to 5] | 3.0 [2 to 4] | 3.0 [1 to 5] | 3.5 [2 to 5] | 3.0 [1 to 5] | 2.0 [1 to 5]
  Texture or Mouth feel Score | 3.0 [1 to 5] | 3.5 [2 to 5] | 2.0 [1 to 4] | 4.0 [1 to 5] | 3.0 [1 to 5] | 4.0 [2 to 5] | 2.0 [1 to 4] | 2.0 [1 to 5]

ADVERSE EVENTS:
Time Frame: From date of first dose of study treatment to date of last dose of study treatment, up to approximately 2 months 10 days
Description: Treatment-emergent adverse events (TEAEs) and serious adverse events were reported. The Safety Analysis Set was the group of subjects who received at least 1 dose of study drug and had at least 1 postdose safety assessment
Arm/Group | Arm 1: 11 mg Lenvatinib Suspension in Water | Arm 1: 11 mg Lenvatinib Capsule With Water | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Juice) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Water) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Juice) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/10 | 0/9 | 0/10 | 0/10 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/10 | 0/9 | 0/10 | 0/10 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 4/19 | 6/20 | 1/10 | 2/9 | 4/10 | 4/10 | 3/18 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 11 mg Lenvatinib Suspension in Water (N=19) | Arm 1: 11 mg Lenvatinib Capsule With Water (N=20) | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Water) (N=10) | Arm 2: 11 mg Lenvatinib (Suspension of 5 Capsules in Juice) (N=9) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Water) (N=10) | Arm 2: 11 mg Lenvatinib (Suspension of 2 Capsules in Juice) (N=10) | Arm 3: 23 mg Lenvatinib Suspension in Water (23 Hours) (N=18) | Arm 3: 23 mg Lenvatinib Suspension in Water (2 Hours) (N=19)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other